CLINICAL TRIAL: NCT05402865
Title: A Real-world Study on Patients of Surgically Unsalvageable or Severe Post-surgery Morbidity Associated Giant Cell Tumor of Bone
Brief Title: A Real-world Study on Patients of Unresectable Giant Cell Tumor of Bone
Status: Completed | Type: Observational
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: JMT103CN03-1
Record Dates: First submitted 2022-05-25; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2021-09

CONDITIONS: Giant Cell Tumor of Bone
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Denosumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Denosumab group: patients who had received denosumab
  Interventions: Drug: Denosumab
- Non-denosumab group: patients who had received anti-GCTB drug therapy other than denosumab, or who did not receive any anti-GCTB medication

INTERVENTIONS:
Drug: Denosumab — Denosumab, subcutaneous injection, specific usage to see the medical records. Non-denosumab, specific usage to see the medical records.
  Other Names: Non-denosumab
  Groups: Denosumab group

SUMMARY:
This is a retrospective observational real-world study, which evaluates the efficacy and safety of denosumab and non-denosumab therapies in the treatment of Chinese populations of surgically unsalvageable or severe post-surgery morbidity associated giant cell tumor of bone (GCTB), collectively referred to as unresectable GCTB, during 2013-2021 in three medical centers, serving as the external control for a single arm phase Ib/II trial on JMT103 treatment of GCTB. 301 patients were enrolled and divided into 2 groups according to their actual previous exposures. Group 1 (n=135) was denosumab group. Group 2 (n=166) included two types of exposures other than denosumab: other anti-GCTB drug therapies, or no therapy on GCTB patients. The dosage, route, frequency and other administration methods was collected according to the actual previous treatment records. The primary outcome measure was the tumor response rate [radiographic tumor response (CR/PR evaluated by ICDs or EORTC criteria) within 12 weeks, or at least 90% reduction of osteoclast like giant cells compared with baseline]. The key secondary endpoint was the tumor response rate [radiographic tumor response (CR/PR evaluated by ICDS or EORTC criteria), or at least 90% reduction of osteoclast like giant cells compared with baseline]. Other secondary Outcome Measures include: proportion of patients whose tumors was surgically resectable; median duration of tumor response (DOR), disease control rate (DCR), and time to disease progression (TTP); and types and proportion of key adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Both genders, aged 18 years or above;
* 2. Patients pathologically diagnosed of giant cell tumor of bone (GCTB), and are surgically unsalvageable, or salvageable but surgery was associated with severe morbidity based on physician's judgement;
* 3. For patients received denosumab or other anti-GCTB medications, one of the two is required: imaging data (including X-ray, CT, MRI or PET-CT) prior to and at least once followed to administration, or pathological data on surgically resected GCTB; for patients with no medication, imaging data or pathological data on surgically resected GCTB is required.

Exclusion Criteria:

* 1. No access to definite treatment information;
* 2. Bone metabolic diseases diagnosed before treatment: hypo-/ hyperparathyroidism, hypo-/hyperthyroidism, hypopituitarism, hyperprolactinemia, Cushing syndrome, acromegaly, Paget disease, etc;
* 3. Complication of malignant tumor receiving anti-tumor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Tumor response rate | 12 weeks (radiology), or through study completion, an average of 1 year (histopathology)
  Radiographic tumor response (CR/PR evaluated by ICDs or EORTC criteria) within 12 weeks, or at least 90% reduction of osteoclast like giant cells compared with baseline

SECONDARY OUTCOMES:
Tumor response rate (Key secondary endpoint) | through study completion, an average of 1 year (radiology and histopathology)
  Radiographic tumor response (CR/PR evaluated by ICDs or EORTC criteria), or at least 90% reduction of osteoclast like giant cells compared with baseline
Proportion of patients that is surgically resectable | through study completion, an average of 1 year
Median duration of tumor response (DOR) | through study completion, an average of 1 year
Disease control rate (DCR) | through study completion, an average of 1 year
Time to disease progression (TTP) | through study completion, an average of 1 year
Types and proportion of key adverse reactions | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - West China Hospital of Sichuan University, Beijing, Beijing Municipality

REFERENCES:
- [Derived] Xu H, Zhou Y, Wei F, Ding Y, Shan H, Yang Y, Liu W, Jin T, Luo Y, Tang F, Lu M, He X, Zhang W, Yang S, Zhang L, Wang J, Li H, Tu C, Niu X. JMT103 versus Non-Denosumab or Denosumab Treatment in Chinese Patients with Unresectable or Surgically Challenging Giant Cell Tumor of Bone: A Propensity Score-Matched Comparison. Cancer Med. 2025 Nov;14(22):e71340. doi: 10.1002/cam4.71340. PMID 41292259